CLINICAL TRIAL: NCT02186171
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Compare the Efficacy and Safety of Romosozumab With Placebo in Men With Osteoporosis
Brief Title: A Study to Compare the Safety and Efficacy of Romosozumab (AMG 785) Versus Placebo in Men With Osteoporosis
Acronym: BRIDGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20110174; 2013-005551-32 (EudraCT Number)
Record Dates: First submitted 2014-06-23; First posted 2014-07-10 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Osteoporosis in Men
Keywords: Osteoporosis in men
MeSH Terms: interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Romosozumab (Experimental): Participants received 210 mg romosozumab administered by subcutaneous injection once a month for 12 months.
  Interventions: Biological: Romosozumab
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injections once a month for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Romosozumab — Administered by subcutaneous injection once a month.
  Other Names: AMG 785; EVENITY™
  Arms: Romosozumab
Drug: Placebo — Administered by subcutaneous injection once a month.
  Arms: Placebo

SUMMARY:
The study is designed to evaluate if treatment with romosozumab once a month for 12 months compared with placebo is effective in increasing bone mineral density (BMD) at the lumbar spine. Additionally, the study will assess the effect of treatment with romosozumab for 12 months compared with placebo on BMD at the femoral neck and total hip.

ELIGIBILITY:
Inclusion Criteria:

* Must be ambulatory male subjects ≥ 55 years to ≤ 90 years of age
* Must have a BMD T score ≤ -2.50 at the spine or hip, or BMD T score ≤ -1.50 at the spine or hip and a history of fragility nonvertebral fracture or vertebral fracture.

Exclusion Criteria:

* A BMD T score ≤ -3.50 at the hip,
* History of hip fracture
* Severe metabolic bone diseases
* Significant laboratory abnormalities
* Recent treatment with agents affecting bone metabolism

Ages: 55 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2016-02-15 (Actual); Study Completion 2016-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (33):
- United States (3):
  - Research Site, Lakewood, Colorado
  - Research Site, Bethesda, Maryland
  - Research Site, Albuquerque, New Mexico
- Belgium (4):
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Colombia (2):
  - Research Site, Medellín, Antioquia
  - Research Site, Bogota, Cundinamarca
- Czechia (3):
  - Research Site, Ostrava-Trebovice
  - Research Site, Pilsen
  - Research Site, Praha 11 - Chodov
- Denmark (2):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
- Japan (7):
  - Research Site, Mizunami-shi, Gifu
  - Research Site, Yokohama, Kanagawa
  - Research Site, Bungoono-shi, Oita Prefecture
  - Research Site, Takatsuki-shi, Osaka
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Toshima-ku, Tokyo
- Mexico (3):
  - Research Site, Mexicali, Baja California Norte
  - Research Site, Monterrey, Nuevo León
  - Research Site, Culiacán, Sinaloa
- Poland (4):
  - Research Site, Lodz
  - Research Site, Świdnik
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Switzerland (2):
  - Research Site, Bern
  - Research Site, Zurich

REFERENCES:
- [Background] Lewiecki EM, Blicharski T, Goemaere S, Lippuner K, Meisner PD, Miller PD, Miyauchi A, Maddox J, Chen L, Horlait S. A Phase III Randomized Placebo-Controlled Trial to Evaluate Efficacy and Safety of Romosozumab in Men With Osteoporosis. J Clin Endocrinol Metab. 2018 Sep 1;103(9):3183-3193. doi: 10.1210/jc.2017-02163. PMID 29931216
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 31 centers in Europe, North America, Latin America, and Japan. Participants were enrolled from 16 June 2014 to 27 January 2015.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive 210 mg romosozumab or matched placebo in a blinded fashion for the duration of the 12-month treatment period. Randomization was stratified by geographic region (Europe, North America, Latin America, and Japan).
Groups:
- Placebo: Participants received placebo subcutaneous injections once a month (QM) for 12 months.
- Romosozumab 210 mg: Participants received 210 mg romosozumab administered by subcutaneous injection once a month for 12 months.
Period: Overall Study
Arm/Group | Placebo | Romosozumab 210 mg
Started | 82 | 163
Received Treatment | 81 | 163
Completed | 78 | 148
Not Completed | 4 | 15
Not completed — Withdrawal by Subject | 1 | 9
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 1 | 2
Not completed — Protocol-specified Criteria | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romosozumab 210 mg | Total
Number analyzed (Participants) | 82 | 163 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (6.9) | 72.4 (7.4) | 72.1 (7.3)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 11 | 31 | 42
  65 - 74 years | 42 | 62 | 104
  75 years and over | 29 | 70 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 82 | 163 | 245
Race [Count of Participants; unit: Participants]
  White | 60 | 120 | 180
  Asian | 9 | 18 | 27
  Black or African American | 0 | 1 | 1
  Other | 13 | 23 | 36
  Multiple | 0 | 1 | 1
Geographic Region [Count of Participants; unit: Participants]
  Europe | 54 | 108 | 162
  Japan | 9 | 18 | 27
  Latin America | 12 | 23 | 35
  North America | 7 | 14 | 21
Lumbar Spine Bone Mineral Density T-score [Mean (Standard Deviation); unit: T-score] — The T-score is the bone mineral density (BMD) at the site when compared to that of a healthy thirty-year-old. Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman.
  T-score | -2.33 (1.41) | -2.22 (1.19) | -2.26 (1.27)
Total Hip BMD T-score [Mean (Standard Deviation); unit: T-score] | -1.92 (0.65) | -1.92 (0.59) | -1.92 (0.61)
Femoral Neck BMD T-score [Mean (Standard Deviation); unit: T-score] | -2.30 (0.52) | -2.34 (0.52) | -2.33 (0.52)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at Month 12
Description: Lumbar spine bone mineral density (BMD) was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline and month 12
Population: Primary efficacy analysis subset, which includes all randomized participants who had a baseline DXA BMD measurement and at least 1 post-baseline DXA BMD measurement at the lumbar spine; last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 210 mg
Number analyzed (Participants) | 79 | 157
percent change | 1.2 (0.5) [lower limit 0.5] | 12.1 (0.5) [lower limit 0.5]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 210 mg; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model adjusting for treatment, baseline BMD value, machine type, machine type-by-baseline BMD value, baseline testosterone level, geographic region, and using a variance structure allowing for heterogeneity between treatment groups; LS Mean Difference = 10.9, 95% CI 2-sided [9.6 to 12.2], Standard Error of Mean 0.6

2. Secondary Outcome: Percent Change From Baseline in BMD at the Total Hip at Month 12
Description: Total hip bone mineral density was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline and month 12
Population: Primary efficacy analysis subset, which includes all randomized participants who had a baseline DXA BMD measurement and at least 1 post-baseline DXA BMD measurement at the total hip; LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 210 mg
Number analyzed (Participants) | 79 | 158
percent change | -0.5 (0.3) [lower limit 0.3] | 2.5 (0.2) [lower limit 0.2]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 210 mg; Test type: Superiority — The Hochberg procedure was employed to control the overall type 1 error for the percent change from baseline at 12 months in total hip and femoral neck to maintain the overall significance level at 0.05; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 3.0, 95% CI 2-sided [2.3 to 3.7], Standard Error of Mean 0.4

3. Secondary Outcome: Percent Change From Baseline in BMD at the Femoral Neck at Month 12
Description: Femoral neck bone mineral density (BMD) was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline and month 12
Population: Primary efficacy analysis subset, which includes all randomized participants who had a baseline DXA BMD measurement and at least 1 post-baseline DXA BMD measurement at the femoral neck; LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 210 mg
Number analyzed (Participants) | 79 | 158
percent change | -0.2 (0.4) [lower limit 0.4] | 2.2 (0.4) [lower limit 0.4]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 210 mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 2.4, 95% CI 2-sided [1.5 to 3.3], Standard Error of Mean 0.5

4. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 6
Description: as for outcome 1
Time Frame: Baseline and month 6
Population: Primary efficacy analysis subset with available data at baseline and month 6.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 210 mg
Number analyzed (Participants) | 78 | 156
percent change | 0.3 (0.4) [lower limit 0.4] | 9.0 (0.4) [lower limit 0.4]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 210 mg; Test type: Superiority — The Hochberg procedure was employed to control the overall type 1 error for the percent change from baseline at 6 months at the lumbar spine, total hip and femoral neck BMD in order to maintain the overall significance level at 0.05; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 8.7, 95% CI 2-sided [7.6 to 9.7], Standard Error of Mean 0.5

5. Secondary Outcome: Percent Change From Baseline in BMD at the Total Hip at Month 6
Description: Bone mineral density was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline and month 6
Population: Primary efficacy analysis subset with available data at baseline and month 6.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 210 mg
Number analyzed (Participants) | 78 | 157
percent change | 0.2 (0.2) [lower limit 0.2] | 1.6 (0.2) [lower limit 0.2]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 210 mg; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 1.4, 95% CI 2-sided [0.8 to 2.0], Standard Error of Mean 0.3

6. Secondary Outcome: Percent Change From Baseline in BMD at the Femoral Neck at Month 6
Description: Bone mineral density (BMD) was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline and month 6
Population: Primary efficacy analysis subset with available data at baseline and month 6.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Romosozumab 210 mg
Number analyzed (Participants) | 78 | 157
percent change | 0.0 (0.4) [lower limit 0.4] | 1.2 (0.3) [lower limit 0.3]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 210 mg; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.0033, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 1.3, 95% CI 2-sided [0.4 to 2.1], Standard Error of Mean 0.4

ADVERSE EVENTS:
Time Frame: 15 months
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Romosozumab 210 mg
Serious Adverse Events (participants affected / at risk) | 10/81 | 23/163
Other Adverse Events (participants affected / at risk) | 41/81 | 74/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Romosozumab 210 mg (N=163)
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 1
Implant site haematoma (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Romosozumab 210 mg (N=163)
Constipation (Gastrointestinal disorders) | 1 | 9
Nasopharyngitis (Infections and infestations) | 22 | 35
Procedural pain (Injury, poisoning and procedural complications) | 6 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 15
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Headache (Nervous system disorders) | 6 | 10
Hypertension (Vascular disorders) | 5 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.